CLINICAL TRIAL: NCT02060266
Title: A Single Centre, Open Label Trial Investigating the Absorption, Metabolism and Excretion After a Single Subcutaneous Dose of [3H]-Semaglutide in Healthy Male Subjects
Brief Title: Trial Investigating the Absorption, Metabolism and Excretion After a Single Subcutaneous Dose of [3H]-Semaglutide in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-3789; 2013-001769-18 (EudraCT Number); U1111-1142-0810 (Other: WHO)
Record Dates: First submitted 2014-02-04; First posted 2014-02-12 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Semaglutide (Experimental)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Subjects will receive a single dose subcutaneously (s.c., under the skin).

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the absorption, metabolism and excretion after a single subcutaneous dose of [3H]-semaglutide in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, based on an assessment of medical history, physical examination, ECG (electrocardiogram) and vital signs, as determined by the investigator
* Age between 45-64 years (both inclusive) at the time of signing inform consent
* Body mass index (BMI) between 20 and 30 kg/m^2 (both inclusive)

Exclusion Criteria:

* Donation of any blood or plasma in the past month or in excess of 100 mL within the 3 months preceding screening, or surgery or trauma with more than 100 mL blood loss within the 3 months preceding screening
* Use of prescription or non-prescription systemic or topical medicinal products (except routine vitamins, acetylsalicylic acid and paracetamol) within 3 weeks (or within 5 half-lives of the medicinal product, whichever is longest) prior to visit 2, Day 1
* History of drug/chemical substance abuse within 1 year from screening, or a positive result in the urine drug test
* History of alcohol abuse within 1 year from screening, or a positive result in the alcohol urine test, or consumption of more than 21 units of alcohol weekly (one unit of alcohol equals about 250 mL of beer or lager, one glass (120 mL) of wine, or 20 mL spirits)
* Smoking or use of any nicotine (including nicotine patches, gum, etc) in the last 3 months prior to screening or a positive nicotine test

Ages: 45 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2014-04-28 (Actual); Study Completion 2014-04-28 (Actual)

PRIMARY OUTCOMES:
Concentration of the major metabolites of [3H]-semaglutide in plasma, urine, and faeces | Up to 9 weeks following a single dose of 0.5 mg [3H]-semaglutide

SECONDARY OUTCOMES:
Total amount of [3H]-semaglutide related material excreted in urine (% of dose) | Up to 9 weeks following a single dose of 0.5 mg [3H]-semaglutide
Total amount of [3H]-semaglutide related material excreted in faeces (% of dose) | Up to 9 weeks following a single dose of 0.5 mg [3H]-semaglutide
Blood to plasma ratio of [3H]-semaglutide related material | Up to 9 weeks following a single dose of 0.5 mg [3H]-semaglutide
Area under the semaglutide plasma concentration curve | From time 0 until infinity after a single dose
Maximum observed semaglutide plasma concentration | After a single dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Groningen, Netherlands

REFERENCES:
- [Result] Jensen L, Helleberg H, Roffel A, van Lier JJ, Bjornsdottir I, Pedersen PJ, Rowe E, Derving Karsbol J, Pedersen ML. Absorption, metabolism and excretion of the GLP-1 analogue semaglutide in humans and nonclinical species. Eur J Pharm Sci. 2017 Jun 15;104:31-41. doi: 10.1016/j.ejps.2017.03.020. Epub 2017 Mar 16. PMID 28323117
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com